CLINICAL TRIAL: NCT02092883
Title: Neuroinflammation in Children With Infantile Spasms Measured With 11C-PK11195 Positron Emission Tomography: Response to ACTH
Brief Title: Evaluation of Neuroinflammation in Children With Infantile Spasms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Harry T Chugani, Professor, Wayne State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 25QNC
Record Dates: First submitted 2014-03-14; First posted 2014-03-20 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Infantile Spasms
Keywords: Infantile Spasms; Neuroinflammation; PK11195; PET; ACTH
MeSH Terms: conditions — Spasms, Infantile; Neuroinflammatory Diseases | interventions — Adrenocorticotropic Hormone

ARMS (1):
- Infantile Spasms (Experimental)
  Interventions: Drug: ACTH

INTERVENTIONS:
Drug: ACTH — PK PET scan before and after ACTH treatment

SUMMARY:
The purpose of this study was to investigate the presence of neuroinflammation in children with infantile spasms using 11C-PK11195 positron emission tomography (PK PET) scan, and its response to ACTH treatment by repeating the PK PET scan after treatment.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of 'cryptogenic IS'
* Normal MRI
* No other neurological disorder

Exclusion Criteria:

* Abnormal MRI
* No anti-inflammatory medication 48 hrs prior to PK PET scans
* Parent/guardian unable to give written consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-03; Primary Completion 2016-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Neuroinflammation in cortical and/or subcortical structures | up to 6 weeks
  Neuroinflammation in cortical and/or subcortical structures of the brain in patients with Infantile Spasms will be evaluated with 11-C-PK11195 PET scan at the baseline and 2 weeks after the completion of ACTH treatment (given over 4 weeks), i.e., 6 weeks after the baseline PET scan.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Michigan, Detroit, Michigan, United States

REFERENCES:
- [Background] Ajay Kumar, Vijay N. Tiwari, Otto Muzik, Pulak K. Chakraborty, Harry T Chugani. In-Vivo Measurement of Brain Inflammation with [11C]-[R]-PK-11195 Positron Emission Tomography in Children with Epileptic Disorders. Epilepsy Currents 2014;14:330 (abs)